CLINICAL TRIAL: NCT06449352
Title: Effect of the Addition of Netarsudil 0.02% vs. Brimonidine 0.1% in Normal Tension Glaucoma Patients Currently on Latanoprost 0.005%
Brief Title: Effect of Netarsudil vs Brimonidine in NTG Patients on Latanoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Westlake Eye Specialists (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ZV-24-01
Record Dates: First submitted 2024-06-03; First posted 2024-06-10 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Normal Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma | interventions — netarsudil; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Netarsudil (Experimental): netarsudil 0.02%
  Interventions: Drug: Netarsudil
- Brimonidine (Active Comparator): brimonidine 0.1%
  Interventions: Drug: Brimonidine

INTERVENTIONS:
Drug: Netarsudil — netarsudil 0.02%
  Arms: Netarsudil
Drug: Brimonidine — brimonidine 0.1%
  Arms: Brimonidine

SUMMARY:
A randomized, multicenter, investigator-masked prospective study of NTG patients currently on latanoprost 0.005% monotherapy, to study the effect of IOP change with the introduction of netarsudil 0.02% vs brimonidine 0.1%. Subjects will be assessed at a screening visit, and 1 follow-up visit. Clinical evaluations will include visual acuity and IOP .

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Diagnosed with normal tension glaucoma based on the following:

  * IOP ≤ 21mmHg
  * Optic nerve rim thinning and/or retinal nerve fiber layer (RNFL) loss consistent with glaucoma
  * Normal visual field OR visual field loss consistent with optic nerve or RNFL defects within the last year
  * Open angles assessed by gonioscopy
* Have been on latanoprost monotherapy for at least 6 weeks

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Patients with angle closure glaucoma or secondary forms of glaucoma due to neovascularization of the angle, uveitic glaucoma, congenital glaucoma, or glaucoma due to congenital anomalies.
* Other forms of secondary glaucoma.
* Patients with abnormal anterior segment examination other than cataract will be excluded from the study.
* Patients who have had incisional surgery for glaucoma (eg: MIGs).
* Patients with refractory CME or CME persisting 3 months or more.
* Children, cognitive impaired and critically ill subjects will not be enrolled.
* Central Corneal Thickness (CCT) ≤ 500.
* Prior allergy to brimonidine or netarsudil, and known to have previously failed either brimonidine or netarsudil.
* Ocular surgery (e.g., cataract, laser, refractive) during the study or 1 year prior to entering the study.

The principal investigator reserves the right to declare a patient ineligible or non- evaluable based on medical evidence that indicates they are unsuitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Mean diurnal intraocular pressure | After 6 weeks of treatment
  Intraocular pressure will be measure at 8am, 12pm, and 4pm

SECONDARY OUTCOMES:
Mean intraocular pressure at 8am | After 6 weeks of treatment
Mean intraocular pressure at 12pm | After 6 weeks of treatment
Mean intraocular pressure at 4pm | After 6 weeks of treatment
Percentage of diurnal intraocular pressure reduction | After 6 weeks of treatment
  Intraocular pressure will be measure at 8am, 12pm, and 4pm

CONTACTS AND LOCATIONS:
Overall Officials: Zarmeena Vendal, MD, Principal Investigator — Westlake Eye Specialists
Locations (4):
- United States (4):
  - Westlake Eye Specialists - Austin Office, Austin, Texas
  - Westlake Eye Specialists - Killeen Office, Killeen, Texas
  - Westlake Eye Specialists - Kyle Office, Kyle, Texas
  - Westlake Eye Specialists - New Braunfels Office, New Braunfels, Texas

IPD SHARING:
Plan to Share IPD: No